CLINICAL TRIAL: NCT05120752
Title: Efficacy of a Low FODMAP Diet in the Absence of Lactose Malabsorption in Moderate to Severe ROME IV IBS.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMaIFI
Record Dates: First submitted 2021-07-13; First posted 2021-11-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FODMAP diet (Experimental)
  Interventions: Other: FODMAP diet

INTERVENTIONS:
Other: FODMAP diet — all participants need to follow a low FODMAP diet, the information will be given by a trained dietitian

SUMMARY:
Irritable bowel syndrome (IBS) is a frequently encountered disorder. According to the Rome IV criteria, it is characterized by abdominal pain associated with a change in stool frequency or con-sistency, or with symptomatic improvement by defecation (Mearin 2016). Associated symptoms, such as bloating and flatulence, are frequently reported. The underlying pathophysiology remains obscure, although several pathways have been proposed. Low-grade immune activation, visceral hypersensitivity, alteration in gut microbiome have all been reported (Mearin 2016). As diet exerts an impact on all these pathophysiological mechanisms, the role of dietary intervention receives spe-cial attention, with special interest in the role played by so-called fermentable oligo-, di-, monosac-charides and polyols (FODMAPs). Multiple studies indicated the beneficial effects of the low FODMAP diet in at least part of the patients (Halmos 2014, Eswaran 2016, Staudacher 2017).

As a disaccharide, lactose is part of the FODMAPs. Lactose intolerance (LI) results from lactose malabsorption (LM) secondary to insufficient hydrolysis of the disaccharide lactose into galactose and glucose (Misselwitz 2019). The undigested lactose will eventually reach the colon, resulting in fermentation from colonic bacteria with production of different compounds such as short chain fat-ty acids, carbon dioxide, H2 and methane (Catanzaro 2021). These compounds have an osmotic effect and can stimulate colonic contractions. In patients suffering from LI, these pathophysiologi-cal mechanisms generate symptoms such as abdominal pain and cramps, flatulence, diarrhea, in-creased bowel sounds, among others, similar to the mechanisms by which FODMAPs induce symp-toms of IBS. As dairy products are highly present in our Western diet, LI will often be considered in patients presenting with such symptoms and they will be referred for further testing. When LM is diagnosed, a lactose-free diet (LFD) will be advocated to alleviate symptoms.

While the earlier-mentioned studies investigated symptomatic improvement by the low FODMAP diet, it remains uncertain whether this restrictive diet remains beneficial in patients without evidence of LM. In a recent study the low FODMAP diet and LFD provided comparable improvement in symptom severity (Krieger-Grübel 2020).

This study aims to:

* Assess the improvement in IBS symptoms and quality of life (QOL) by a low FODMAP di-et when lactose malabsorption has been previously excluded;
* Compare the improvement in IBS symptoms and QOL obtained by a low FODMAP diet to a lactose free diet (data from the PreVaIL study).

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged 18 - 75 years;
* Fulfilling the ROME IV criteria for IBS;
* Moderate symptom severity as defined by a IBS-SSS > 175;
* Consumption of lactose containing products.

Exclusion Criteria:

* - Clinical suspicion of an organic disorder different from LI or IBS (patients can be included when this disorder had been excluded);
* Known lactose intolerance;
* Known inflammatory bowel disorder;
* Known major intestinal motility disorder;
* Alcohol (defined as more than 14 U per week) or other substance abuse;
* Active psychiatric disorder;
* Known systemic or auto-immune disorder with implication for the GI system;
* Prior abdominal surgery (with the exception of appendectomy);
* Any prior diagnosis of cancer other than basocellular carcinoma;
* Current chemotherapy;
* History of gastro-enteritis in the past 8 weeks;
* Intake of antibiotics, pre- or probiotics during the past 8 weeks;
* Dietary supplements unless taken at a stable dose for more than 8 weeks;
* Treatment with neuromodulators (one neuromodulator taken at a stable dose for more than 12 weeks is allowed);
* Treatment with spasmolytic agents, opioids, loperamide, gelatin tannate or mucoprotectants during the past 8 weeks;
* LFD or low FODMAP diet in the past.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
symptomatic improvement | 3 to 4 months
  To evaluate the symptomatic improvement by a low FODMAP diet in Rome IV IBS patients with-out documented lactose malabsorption.
Evolution of Quality of life scale | 3 to 4 months
  Evolution of quality of life by the low FODMAP diet.

SECONDARY OUTCOMES:
reduction in Irritable bowel syndrome - symptom severity scale | baseline till week 4, baseline till week 16
  Reduction of IBS-SSS at 4 weeks of diet vs. baseline depending on the reduction of FOD-MAP consumption;

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Kindt, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No